CLINICAL TRIAL: NCT05261789
Title: Comparison of the Effects of Turkish Get Up Exercise and Stabilization Exercises on Muscular Activation, Core Stability and Upper Extremity Performance in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-168
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Physical Therapy
Keywords: Exercise; Core Stability; Upper Extremity Performance
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Including healthy male individuals between the ages of 18-25. The participants will randomly be allocated three groups (TGU exercise group, core stability exercise group and control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Turkish Get Up exercise group (Experimental): Turkish Get Up exercise was given this group
  Interventions: Other: Turkish Get Up exercise
- Core stability exercise group (Experimental): Core stability exercise was given this group
  Interventions: Other: Core Stability exercise
- Control group (Active Comparator): No intervention
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Turkish Get Up exercise — Before the exercise, warm-up exercises (low intensity aerobic activity, short-term stretches) were applied for 5 minutes. 7 different steps (1. Starting position, 2. Supine kettlebell lift, 3. Elbow-supported kettlebell lift, 4. Hand-supported kettlebell lift, 5. High bridge, 6. Half-kneeling and lunge position, 7. Standing up) and the return of these different steps, a total of 2 stages exercise program was applied.
  The exercise was started with 3 repetitions for each side and 3 sets with a 30-second rest period between repetitions, and 2 minutes of rest between sets. At the beginning of the 3rd week, the exercise was applied as 3 sets of 4 repetitions, and at the beginning of the 5th week, 3 sets of 5 repetitions were applied. At the end of the exercise, cool-down exercises (low intensity jogging and static stretching) were applied for 5 minutes.
  Arms: Turkish Get Up exercise group
Other: Core Stability exercise — After the individuals were taught how to activate their core muscles before the exercise, they were asked to do bridge, prone and lateral bridge exercises by contracting their core muscles. Before the exercises, warm-up exercises (low intensity aerobic activity, short-term stretches) were applied for 5 minutes.
  Bridge exercise, prone bridge exercise, lateral bridge exercise were applied
  Arms: Core stability exercise group
Other: Control Group — No exercise will be applied to the individuals in the control group. At the end of the 6-week period, all parameters will be evaluated again.
  Arms: Control group

SUMMARY:
Turkish Get Up (TGU) exercise, which is one of the kettlebell exercises, is a multi-step, progression-based, functional and whole-body exercise method that includes a combination of movements such as lunge, bridge building and side plank. Strength training, dynamic flexibility exercises and strength training can be performed with the use of a kettlebell. Exercises with a kettlebell are frequently used in the fields of improving sportive performance and rehabilitation. TGU exercise can be used as a corrective exercise as well as in motion analysis and conditioning studies. TGU exercise consists of 2 stages:The first stage is performed in seven different steps: 1. Starting position, 2. Supine kettlebell lift, 3. Elbow-supported kettlebell lift, 4. Hand-supported kettlebell lift, 5. High bridge, 6. Half-kneeling and lunge position, 7. Stand up. In the second stage, the exercise is completed by performing the return of the steps in the first stage. It is thought that the deltoid, rectus abdominis, external oblique abdominis, erector spinae, gluteal muscles, quadriceps and hamstring muscles are activated during this exercise. It has been reported that with the TGU exercise, especially rotator cuff muscle strength, shoulder stability, balance and core stability can be improved.

In the literature, there are many studies examining the effects of stabilization exercises on core muscles. On the other hand, although there are studies reporting that the TGU exercise can improve core stability and shoulder stability, and studies reporting the muscular activation of the shoulder girdle muscles and some trunk muscles during the TGU exercise. To the best of our knowledge, we have not found a study examining its effectiveness on muscle activation, core stability and upper extremity performance and comparing it with any other method.

The aim of this study is to compare the effects of TGU exercise and stabilization exercises on muscular activation, core stability and upper extremity performance in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male individuals, between the ages of 18-25, Individuals whose physical activity levels are at least 3000 MET min/week and above according to the International Physical Activity Questionnaire-Short Form, Individuals with a body mass index of 17-30 kg/m2

Exclusion Criteria:

* Professionally engaged in sports, Have any known orthopedic, neurological or cardiovascular problems, Having undergone musculoskeletal surgery in the last 1 year, Individuals who have had a musculoskeletal injury in the last 3 months.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Core stability | 6 weeks
  Core stability of individuals, static endurance; were performed with trunk flexors endurance test, Measurement were recorded in seconds using a digital stopwatch.
Core stability | 6 weeks
  Core stability of individuals, static endurance; were performed with trunk extensors endurance test, Measurement were recorded in seconds using a digital stopwatch.
Core stability | 6 weeks
  Core stability of individuals, static endurance; were performed with lateral bridge endurance test, Measurement were recorded in seconds using a digital stopwatch.
Core stability | 6 weeks
  Core stability of individuals, static endurance; were performed with the prone bridge test, Measurement were recorded in seconds using a digital stopwatch.
Muscle activation | 6 weeks
  Muscle activations of individuals were evaluated using superficial EMG. An 8-channel EMG Noraxon MiniDTS system (Noraxon, USA, Inc, Scottsdale, AZ) was used to measure signals from the muscles. Before placing the electrodes, the skin was prepared by shaving the area to be treated and cleaning with alcohol cotton until the skin was slightly red in order to reduce the skin impedance. Electrodes, Surface It was placed parallel to the muscle fibers at the points recommended by ElectroMyoGraphy for the Non-Invasive Assessments of Muscles (SENIAM). On the dominant side of individuals; Electrodes were placed 15 cm lateral to the umbilicus for external oblique abdominis, 2 cm above and 3 cm lateral to the umbilicus for rectus abdominis, and 3 cm lateral to the L3 spinous process for lumbar erector spinae.
Upper extremity performance | 6 weeks
  The upper extremity Y balance test was used to evaluate the balance, function and stability of the upper extremity and trunk. In the initial phase of the test, the individual took a push-up position with arms shoulder-width apart. Before the test, the individual was allowed to try 3 times for warming up. During the test phase, the nondominant hand was extended 3 times in the medial, inferior lateral and superior lateral directions, and the distance was recorded, and then the dominant hand was passed. Composite score was obtained by dividing the total score of 3-repetition distance for each direction by 3 times the length of the upper extremity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No